CLINICAL TRIAL: NCT07045961
Title: Concurrent Exercise in Combination With Music Listening in Female Breast Cancer Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ana Trigueros Murillo (Other)
Responsible Party: Sponsor-Investigator, Ana Trigueros Murillo, MSc, Physiotherapy, University of Seville
Organization: University of Seville (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-0855
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Survivors
Keywords: Breast cancer survivors; Concurrent exercise; Music medicine; Randomized controlled trial

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, parallel assignment. Participants will be equally assigned (1:1) to one of two groups. The experimental group will receive a concurrent exercise program (combining strength and endurance training) enhanced with music medicine. The control group will undergo the same concurrent exercise program without music therapy, serving as an active comparator.The evaluator will remain blinded to the intervention assigned to each participant throughout the study .
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent Exercise and Music Medicine (Experimental): Supervised Station-Based Strength Circuit Training (2 sessions/week) combined with music medicine.
  Interventions: Other: Supervised Station-Based Strength Circuit Training & Self-directed aerobic training; Other: Music Medicine
- Concurrent exercise (Active Comparator): Supervised Station-Based Strength Circuit Training (2 sessions/week)
  Interventions: Other: Supervised Station-Based Strength Circuit Training & Self-directed aerobic training

INTERVENTIONS:
Other: Supervised Station-Based Strength Circuit Training & Self-directed aerobic training — Anaerobic training sessions follow a circuit design alternating upper body, lower body, and core exercises with dumbbells, barbells, and kettlebells. Participants complete 3 sets of 10-15 repetitions per exercise, performed consecutively without rest, at 60-80% of their one-repetition maximum (1RM). Two participants perform the same exercise simultaneously at each station. Load progression is applied by increasing resistance by 10% after successfully completing 3 sets of 12 repetitions across two consecutive sessions.
  Sessions begin with a 5-minute warm-up at 50-65% of maximal heart rate (HRmax), followed by nine resistance exercises: kettlebell squats, static plank, bench press, weighted lunges, quadruped superman, seated row, weighted glute bridge, leg raises, and shoulder press. Exercises alternate muscle groups to optimize recovery.
  Additionally, participants engage in self-selected aerobic exercise (walking, running, rowing, swimming, or stationary cycling) twice weekly at 65-80
Other: Music Medicine — During the warm-up phase, participants will engage in individual passive music listening, tailored to their personal musical preferences. The music will be delivered via MP3 players or smartphones, where a personalized playlist containing the participant's favorite tracks has been preloaded. Subsequently, during the circuit training session, a group background music playlist will be played through speakers. This heterogeneous playlist is compiled based on the collective musical preferences of all participants. Finally, during the cool-down phase, a common background music selection will be used, featuring a different repertoire from earlier phases. The cool-down will include guided muscle relaxation and breathing exercises assisted by the background music.
  Arms: Concurrent Exercise and Music Medicine

SUMMARY:
This clinical trial aims to compare the effects of a concurrent physical exercise program (aerobic and resistance training) combined with music medicine versus exercise alone on self-perception (self-esteem and body image), physical condition (strength, fatigue, cardiovascular endurance) and general well-being (quality of life and sleep quality) in female breast cancer survivors.

The main research question is:

- Is a program that combines physical exercise and music therapy more effective than physical exercise alone in improving self-perception, physical condition, and general well-being in breast cancer survivors?

Participants will be randomly assigned to one of two groups:

* One group will receive concurrent physical exercise combined with music therapy.
* The other group will receive the same exercise program without music therapy. Assessments will be conducted at three time points: before the intervention, immediately after the intervention, and 6 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 75 years with a prior diagnosis of stage 0-III breast cancer.
* Women currently in the survivorship phase of the disease, regardless of the type of medical or surgical treatment received.
* A minimum of six months must have elapsed since the completion of primary treatment.

Exclusion Criteria:

* History of lymphedema secondary to axillary surgery.
* Inability to provide informed consent for participation in the study.
* Prior diagnosis of hearing impairments that hinder or prevent music listening, such as partial or total deafness.
* Prior diagnosis of any central or peripheral neurological condition.
* Presence of comorbidities or conditions that contraindicate participation in a physical exercise program.

  * A preliminary screening of participants will be conducted based on the recommendations of the National Comprehensive Cancer Network (NCCN), considering the risk of potential exercise-induced adverse effects.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Self-Esteem Measured by the Rosenberg Self-Esteem Scale (RSES). | Self-esteem will be assessed at three time points: prior to the intervention (baseline), immediately following the intervention (post-intervention), and at 6-month follow-up.
  The instrument evaluates constructs of self-worth and self-acceptance via 10 items, comprising five positively phrased and five negatively phrased statements, each scored on a 4-point Likert scale (1 = strongly agree, 2 = agree, 3 = disagree, 4 = strongly disagree). Total scores range from 10 to 40 points, with reverse scoring applied to negatively worded items to ensure accurate assessment. Elevated total scores correspond to higher self-esteem levels. The scale exhibits robust internal consistency (Cronbach's alpha = 0.87) and established construct validity

SECONDARY OUTCOMES:
Change from Baseline in Body Image Measured by the Hopwood Body Image Scale (S-BIS). | Body image will be assessed at three time points: prior to the intervention (baseline), immediately following the intervention (post-intervention), and at 6-month follow-up.
  The S-BIS is a psychometrically validated instrument comprising 10 items that assess multiple dimensions of body image, including affective, cognitive, and behavioral domains. Responses are recorded on a 4-point Likert scale ranging from 0 (not at all) to 3 (very much). Total scores span from 0 to 30, with elevated scores (21-30) indicative of pronounced disturbances in body image perception. The scale exhibits excellent internal consistency reliability (Cronbach's alpha = 0.966).
Change from Baseline in Fatigue Levels Measured by the Piper Fatigue Scale (PFS). | Fatigue will be assessed at three time points: prior to the intervention (baseline), immediately following the intervention (post-intervention), and at 6-month follow-up.
  The Piper Fatigue Scale is a 22-item questionnaire scored from 0 to 10 that assesses behavioral, affective, sensory, and cognitive dimensions of fatigue. The maximum score, indicating high levels of fatigue, is 220 points. The instrument demonstrates good internal consistency, with a Cronbach's alpha greater than 0.86. Construct and criterion validity have been established
Change from Baseline in Upper Limb Strength Measured by Handgrip Dynamometry. | Handgrip strength will be assessed at three time points: prior to the intervention (baseline), immediately following the intervention (post-intervention), and at 6-month follow-up.
  A handgrip dynamometer will be used to assess grip strength with the patient in a standing position and the elbow flexed at 90°. The test will be performed alternately three times on each hand, with a one-minute rest interval between trials. Higher kilogram values correspond to greater grip strength. This procedure is considered the gold standard for assessing upper limb strength.
Change from Baseline in Lower Limb Strength Measured by the 5-Repetition Sit-to-Stand Test (5STS). | Handgrip strength will be assessed at three time points: prior to the intervention (baseline), immediately following the intervention (post-intervention), and at 6-month follow-up.
  This is a functional test designed to assess lower limb strength. Participants begin the test seated on an armless chair with a seat height between 41 and 45 cm, with their arms crossed over the chest. They are instructed to stand up and sit down five times consecutively as quickly as possible without using their upper limbs for support. Timing is recorded with a stopwatch, starting at the verbal cue 'go' and stopping when the participant sits after the fifth repetition. Longer completion times may indicate muscle weakness.
Change from Baseline in Cardiovascular Endurance Measured by the 6-Minute Walk Test (6MWT). | Cardiovascular endurance will be assessed at three time points: prior to the intervention (baseline), immediately following the intervention (post-intervention), and at 6-month follow-up.
  This test evaluates physical and Cardiovascular endurance calculating the maximum distance the participant is able to walk over six minutes on a predefined course set along a flat indoor corridor with two turning points. Longer walking distances reflect superior cardiovascular and functional aerobic capacity. Its reliability and validity in patients with cancer have been demonstrated, with an intraclass correlation coefficient (ICC) of 0.93.
Change from Baseline in Quality of Life Measured by the Functional Assessment of Cancer Therapy-Breast (FACT-B), Version 4. | Quality of Life will be assessed at three time points: prior to the intervention (baseline), immediately following the intervention (post-intervention), and at 6-month follow-up.
  This 37-item questionnaire comprises four subscales assessing physical, social/family, emotional, and functional well-being, along with a breast cancer-specific domain. Items are rated on a 5-point Likert scale (0 = not at all; 4 = very much), with a maximum total score of 148 points. Higher scores indicate better quality of life. The instrument demonstrates high overall internal consistency (Cronbach's alpha = 0.90), and its validity and test-retest reliability have been confirmed.
Change from Baseline in Sleep Quality Measured by the Pittsburgh Sleep Quality Index (PSQI) | Handgrip strength will be assessed at three time points: prior to the intervention (baseline), immediately following the intervention (post-intervention), and at 6-month follow-up.
  The questionnaire is structured into seven major components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is rated on a scale from 0 (no difficulty) to 3 (severe difficulty), based on patient-reported data. A global score of 0 reflects no sleep difficulties, whereas the maximum score of 21 indicates extreme sleep impairment. The index demonstrates moderate-to-high internal consistency (Cronbach's alpha = 0.81) in clinical populations. Its criterion validity shows a sensitivity of 90% and a kappa index of 0.6.

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Physiotherapy and Podiatry, Faculty of Nursing, Physiotherapy and Podiatry, University of Seville, Spain (Avicena Street, s/n), Seville, España, Spain

REFERENCES:
- See also: National Comprehensive Cancer Network (NCCN) — https://bmtinfonet.org/es/resource/red-nacional-integral-del-cancer-national-comprehensive-cancer-network